CLINICAL TRIAL: NCT00792701
Title: Phase II ERCC1 and RRM1-Based Adjuvant Therapy Trial in Patients With Stage I Non-Small Cell Lung Cancer (NSCLC)
Brief Title: S0720: Adjuvant Therapy Based on Gene Expression in Stage IA and IB Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000625070; S0720 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2008-11-16; First posted 2008-11-18 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm II (Experimental): Beginning within 84 days after surgery, patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and cisplatin IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cisplatin; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: cisplatin — Given IV
Drug: gemcitabine hydrochloride — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy drugs after surgery may kill any tumor cells that remain after surgery. Sometimes, after surgery, the tumor may not need more treatment until it progresses. In this case, observation may be sufficient.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with cisplatin works in treating patients with stage I non-small cell lung cancer that was removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the feasibility of assigning adjuvant treatment based on tumoral RRM1 and ERCC1 gene expression in patients with complete surgical resection of stage IA (≥ 2 cm) or IB non-small cell lung cancer.

Secondary

* To estimate the collective 2-year disease-free survival of these patients.
* To assess the frequency and severity of toxicities resulting from the administration of cisplatin and gemcitabine hydrochloride.
* To explore, preliminarily, the relationship between RNA and protein expression of RRM1 and ERCC1, and the relationship between RRM1 and ERCC1 expression in the formalin-fixed and paraffin-embedded tumor specimens, and to generate results on in situ protein expression and other assays for genes involved in drug efficacy.
* To assess the analytical performance of the biomarker assay.

OUTLINE: This is a multicenter study.

Patients are assigned to 1 of 2 treatment arms based on RRM1 and ERCC1 gene expression.

* Arm I (RRM1 ≥ 40 and ERCC1 ≥ 65): Patients undergo active monitoring after surgery with disease assessments at 8, 16, and 24 weeks.
* Arm II (RRM1 < 40 and/or ERCC1 < 65): Beginning within 84 days after surgery, patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and cisplatin IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Tumor samples acquired at the time of surgery are analyzed by immunofluorescence-based automated quantitative analysis for in situ expression of RRM1 and ERCC1. If available, additional samples are assessed using RT-PCR and real-time quantitative PCR for RRM1 and ERCC1 expression levels; polymorphism analysis for RRM1 and ERCC1 expression at the protein level; and tissue microarray analysis of genes associated with DNA synthesis, damage repair, and drug efficacy.

After completion of study therapy, patients are followed every 6 months for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer

  * Stage IA (longest tumor diameter 2-3 cm) or stage IB disease
* Must have undergone preoperative CT scan of the chest (including the entire liver and adrenals) with IV contrast AND a whole body PET scan or a combined PET/CT scan with no evidence of N1, N2, N3, or M1 disease within 42 days prior to surgery
* A whole body PET scan or a combined PET/CT must be performed within 84 days

  * Any finding on PET scan that clinically suggests N1, N2, N3, or M1 disease must have been cleared by further evaluation, including, but not limited to, any of the following:

    * Ultrasonography, X-ray radiology, magnetic resonance imaging, or nuclear medicine imaging
* Completely resected (R0) disease by lobectomy, bilobectomy, or pneumonectomy performed by open thoracotomy or video-assisted thoracoscopic surgery within the past 35 days

  * Completely excised primary lesion with negative gross and microscopic margins
  * At least two mediastinal lymph node stations sampled
* Must have tumor tissue available from the surgical resection specimen AND agree to have treatment assignment determined by a gene expression analysis performed on that tissue

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 mg/dL
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 1.5 times ULN
* Serum creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior malignancy except for the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated stage I-II cancer from which the patient is currently in complete remission
  * Any other cancer from which the patient has been disease-free for 5 years
* Willing to provide prior smoking history

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior systemic chemotherapy or biologic therapy for lung cancer
* No prior thoracic radiation therapy (RT) (including RT to the chest wall)
* No other concurrent investigational agents, chemotherapeutic agents, RT, or hormonal therapy

  * Steroids administered for antiemesis, adrenal failure, or septic shock OR hormones administered for non-disease-related conditions (e.g., insulin for diabetes) allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2008-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph G. Zinner, MD, Study Chair — M.D. Anderson Cancer Center
Locations (147):
- United States (147):
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Sherman Hospital, Elgin, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Caritas St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - AnMed Cancer Center, Anderson, South Carolina
  - Cancer Centers of the Carolinas - Easley, Easley, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Eastside, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Self Regional Cancer Center at Self Regional Medical Center, Greenwood, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Greer Radiation Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Northwest Cancer Specialists at Vancouver Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Derived] Bepler G, Zinner RG, Moon J, Calhoun R, Kernstine K, Williams CC, Mack PC, Oliveira V, Zheng Z, Stella PJ, Redman MW, Gandara DR. A phase 2 cooperative group adjuvant trial using a biomarker-based decision algorithm in patients with stage I non-small cell lung cancer (SWOG-0720, NCT00792701). Cancer. 2014 Aug 1;120(15):2343-51. doi: 10.1002/cncr.28714. Epub 2014 Apr 18. PMID 24752945

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Monitoring: Patients undergo active monitoring after surgery with disease assessments at 8, 16, and 24 weeks.
  Active surveillance: Patients undergo active monitoring
- Gemcitabine Hydrochloride and Cisplatin: Beginning within 84 days after surgery, patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and cisplatin IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Cisplatin: Given IV
  Gemcitabine Hydrochloride: Given IV
Period: Overall Study
Arm/Group | Active Monitoring | Gemcitabine Hydrochloride and Cisplatin
Started | 19 | 66
Eligible | 18 | 63
Eligible and Analyzable | 17 | 44
Completed | 0 | 22
Not Completed | 19 | 44
Not completed — Adverse Event | 0 | 22
Not completed — Ineligible | 1 | 3
Not completed — Withdrawal by Subject | 1 | 19
Not completed — Not protocol specified | 17 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Monitoring | Gemcitabine Hydrochloride and Cisplatin | Total
Number analyzed (Participants) | 18 | 63 | 81
Age, Continuous [Median (Full Range); unit: years] | 68.8 [41.6 to 81.7] | 63.3 [41.6 to 84.2] | 64 [41.6 to 84.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 37 | 44
  Male | 11 | 26 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 58 | 74
  Unknown or Not Reported | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 0 | 8 | 8
  White | 14 | 52 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 8 | 44 | 52
  Squamous | 8 | 17 | 25
  Large Cell | 0 | 1 | 1
  Bronchioloalveolar | 1 | 0 | 1
  Other | 1 | 1 | 2
Performance Status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  3. Capable of limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled; cannot carry on any self-care; totally confined to bed or chair.
  Participants
    0 | 13 | 31 | 44
    1 | 5 | 32 | 37
Smoking History [Count of Participants; unit: Participants]
  Current | 7 | 26 | 33
  Former | 9 | 30 | 39
  Never | 2 | 7 | 9
Stage [Count of Participants; unit: Participants] — At the time of surgery, patients must have Stage IA (with the longest tumor diameter ≥ 2 cm) or Stage IB disease as outlined below (AJCC Cancer Staging Manual, 6th Edition, 2002):
  Stage IA (with longest tumor diameter ≥ 2 cm)
  * T1
  * N0
  * M0
  Stage IB
  * T2
  * N0
  * M0
  Participants
    IA | 3 | 22 | 25
    IB | 15 | 41 | 56
Weight Loss Last 6 Months [Count of Participants; unit: Participants]
  <5% | 15 | 49 | 64
  5-<10% | 2 | 7 | 9
  10-20% | 1 | 3 | 4
  >20% | 0 | 1 | 1
  Unknown | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Pharmacogenomics-based Treatment Assignment in the Cooperative Group Setting
Description: Feasibility will be assessed both by accrual rate and the percentage of patients successfully assigned to adjuvant chemotherapy or active monitoring.
Time Frame: From time of registration to 84 days after surgical resection.
Population: Percentage of patients successfully assigned to adjuvant chemotherapy or active monitoring.
Measure: Count of Participants; unit: Participants
Groups:
- All Eligible Patients: All patients who received a treatment assignment within the prespecified timeframe.
Arm/Group | All Eligible Patients
Number analyzed (Participants) | 81
Participants | 71

2. Secondary Outcome: Two-year Disease-free Survival
Time Frame: From time of registration to maximum of 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Active Monitoring | Gemcitabine Hydrochloride and Cisplatin
Number analyzed (Participants) | 17 | 44
percentage of participants | 71 [43 to 87] | 83 [68 to 91]

3. Secondary Outcome: Frequency and Severity of Toxicities as Assessed by NCI CTCAE v3.0
Description: Patients in the active monitoring arm were not followed for adverse events.
Time Frame: From time of registration to maximum of 2 years
Population: Number of Subjects With Greater Than Grade 2 Toxicity
  Patients in the active monitoring arm were not followed for adverse events.
Measure: Number; unit: participants
Arm/Group | Gemcitabine Hydrochloride and Cisplatin
Number analyzed (Participants) | 43
participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 1
  Anorexia | 2
  Dehydration | 1
  Fatigue (asthenia, lethargy, malaise) | 2
  Febrile neutropenia | 2
  Hearing: pts w/o audiogram not enroll monitor prgm | 1
  Hemoglobin | 2
  Mucositis/stomatitis (clinical exam) - Oral cavity | 1
  Nausea | 4
  Neutrophils/granulocytes (ANC/AGC) | 17
  Platelets | 8
  Pleural effusion (non-malignant) | 1
  Potassium, serum-low (hypokalemia) | 1
  Renal failure | 1
  SVT and nodal arrhythmia - Sinus bradycardia | 1
  Sodium, serum-low (hyponatremia) | 2
  Syncope (fainting) | 1
  Thrombosis/embolism (vascular access-related) | 1
  Thrombosis/thrombus/embolism | 1
  Vomiting | 4

4. Secondary Outcome: Relationship Between RRM1 and ERCC1 Expression in the Formalin-fixed and Paraffin-embedded Tumor Specimens.
Description: RRM1 and ERCC1 protein levels are expressed as a simple score with no units.
Time Frame: From time of registration to maximum of 2 years
Population: Protein expression relationships were analyzed in the overall patient population, and not by arm.
Measure: Median (Full Range); unit: Scores
Groups:
- All Patients: All registered patients.
Arm/Group | All Patients
Number analyzed (Participants) | 85
Scores
  RRM1 Protein Score | 39.7 [2.4 to 234.3]
  ERCC1 Protein Score | 41.9 [4.3 to 211.2]
Statistical Analysis 1: Comparison: All Patients; Test type: Other — Correlation; p = 0.003, t-test, 2 sided; Correlation Coefficient = 0.39

5. Other Pre Specified Outcome: Analytical Performance of the Biomarker Assay
Time Frame: From time of registration to maximum of 2 years
Population: Due to lack of funding, the assay was never performed. Thus, this outcome could not be analyzed.
Arm/Group | All Patients
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Generation of Results on in Situ Protein Expression and Other Assays for Genes Involved in Drug Efficacy
Time Frame: From time of registration to maximum of 2 years
Population: Due to lack of funding, the protein expression data were never collected. Thus, this outcome could not be analyzed.
Arm/Group | All Patients
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Relationship Between RNA and Protein Expression of RRM1 and ERCC1
Time Frame: From time of registration to maximum of 2 years
Measure: Median (Full Range); unit: Scores
Arm/Group | All Patients
Number analyzed (Participants) | 81
Scores
  RRM1 Protein Score | 39.7 [2.4 to 234.3]
  ERCC1 Protein Score | 41.9 [4.3 to 211.2]
Statistical Analysis 1: Comparison: All Patients; Comparing RRM1 levels and ERCC1 levels between all patients; Test type: Superiority or Other; p = .0003, Chi-squared; Correlation Coefficient = .39

ADVERSE EVENTS:
Time Frame: From time of registration to maximum of 2 years. Patients in the active monitoring arm were not followed for adverse events.
Description: All SAEs and AEs
  Patients in the active monitoring arm were not followed for adverse events.
Groups:
- Gemcitabine Hydrochloride and Cisplatin: Beginning within 84 days after surgery, patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and cisplatin IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Gemcitabine Hydrochloride and Cisplatin
Serious Adverse Events (participants affected / at risk) | 2/43
Other Adverse Events (participants affected / at risk) | 41/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine Hydrochloride and Cisplatin (N=43)
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine Hydrochloride and Cisplatin (N=43)
Hemoglobin (Blood and lymphatic system disorders) | 25
Tinnitus (Ear and labyrinth disorders) | 12
Constipation (Gastrointestinal disorders) | 16
Diarrhea (Gastrointestinal disorders) | 10
Heartburn/dyspepsia (Gastrointestinal disorders) | 6
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 4
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 34
Vomiting (Gastrointestinal disorders) | 18
Edema: limb (General disorders) | 6
Fatigue (asthenia, lethargy, malaise) (General disorders) | 31
Pain-Other (General disorders) | 3
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 6
AST, SGOT (Investigations) | 10
Alkaline phosphatase (Investigations) | 9
Creatinine (Investigations) | 3
Leukocytes (total WBC) (Investigations) | 12
Metabolic/Laboratory-Other (Investigations) | 4
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 28
Platelets (Investigations) | 14
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 18
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 6
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 15
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 3
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 6
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 8
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 4
Pain - Back (Musculoskeletal and connective tissue disorders) | 4
Pain - Joint (Musculoskeletal and connective tissue disorders) | 4
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 13
Neuropathy: sensory (Nervous system disorders) | 7
Pain - Head/headache (Nervous system disorders) | 12
Taste alteration (dysgeusia) (Nervous system disorders) | 10
Insomnia (Psychiatric disorders) | 10
Mood alteration - anxiety (Psychiatric disorders) | 5
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 3
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 7
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 4
Thrombosis/thrombus/embolism (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No